CLINICAL TRIAL: NCT00879112
Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy, Safety, and Tolerability of MB07811 for 12 Weeks Followed by a 6-Week Off Drug Phase in Subjects With Primary Hypercholesterolemia
Brief Title: Study of MB07811 in Subjects With Hypercholesterolemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated prior to initiation
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Director, Project Management, Ligand Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB07811-201
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — 2-((3,5-dimethyl-4-(4'-hydroxy-3'-isopropylbenzyl)phenoxy)methyl)-4-(3-chlorophenyl)-2-oxido(1,3,2)dioxaphosphonane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): MB07811 Cohort 1
  Interventions: Drug: MB07811
- 2 (Experimental): MB07811 Cohort 2
  Interventions: Drug: MB07811
- 3 (Experimental): MB07811 Cohort 3
  Interventions: Drug: MB07811
- 4 (Placebo Comparator): Cohort 4
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MB07811 — Oral
  Arms: 1; 2; 3
Drug: Placebo — Oral
  Arms: 4

SUMMARY:
A Phase 2 randomized, placebo controlled study assessing the efficacy, safety, and tolerability of MB07811 given orally to subjects with primary hypercholesterolemia for 12 weeks followed by a 6-week off drug phase.

DETAILED DESCRIPTION:
This is an outpatient, Phase 2, multicenter, double-blind, placebo-controlled, randomized, parallel-group study assessing the efficacy, safety, and tolerability of MB07811 given orally to subjects with primary hypercholesterolemia for 12 weeks. There will be a 3- to 6-week screening/run-in period, including washout of any lipid-modifying therapies (as needed) prior to randomization. Eligible subjects will be randomized (1:1:1:1) to placebo, or 3 different doses of MB07811 for 12 weeks. After the double-blind treatment phase, all randomized subjects will proceed into a 6-week off-drug phase. Assessments include: laboratory tests, adverse events (AEs), electrocardiograms (ECGs), vitals, and PK samples.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18.50 - 40 kg/m2 inclusive at screening;
* Fasting serum LDL-C ≥145 mg/dL at both Q2 and Q3 visits;
* Fasting mean serum LDL-C <220 mg/dL from Q2 and Q3;

Exclusion Criteria:

* History of clinically significant cardiovascular disease
* Uncontrolled hypertension
* Significant sinus bradycardia defined as <40 beats per minute (bpm);
* Personal or family history of clinically significant unexplained syncope, near-syncope or unexplained sudden death or QT syndrome;
* Holter monitor report demonstrating any abnormality that is clinically significant, including but not limited to PVC frequency > 1 per minute, any alert criteria or any other condition that requires further evaluation;
* History of clinical significant arrhythmia;
* Resting 12-lead ECG showing QTc >450 msec or <360 msec (males or females), any tachyarrhythmia or morphology change, or any other clinically significant abnormality;
* Any other cardiovascular event requiring hospitalization;
* History or presence of thyroid disorder or other metabolic/endocrine disorder that affects lipids or glucose; Exceptions: polycystic ovarian syndrome (PCOS) and impaired glucose tolerance (IGT) are allowed.
* Liver disease, gallbladder disease, Gilbert's syndrome, biopsy-proven nonalcoholic steatohepatitis (NASH), positive serology for hepatitis B surface antigen (HBsAg) or hepatitis C antibodies; Exceptions: gallbladder disease treated with cholecystectomy
* History of human immunodeficiency virus (HIV);
* Subjects with a prior history of malignancy in past 5 years;Exceptions: Subjects with previous history of basal or squamous cell carcinoma of the skin, or cervical cancer in situ are allowed if successfully treated;
* History of myopathy, including any history of statin-induced myopathy;
* History of intolerance to statins (e.g., myalgias, elevated liver tests);
* History of clinically significant psychiatric disorders, including but not limited to bipolar disorder, major depressive disorder, psychosis;
* Renal dysfunction;
* Alcohol and/or drug abuse within 12 months prior to screening;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effects of MB07811 compared to placebo on LDL-C | 12-weeks of treatment

SECONDARY OUTCOMES:
Evaluate the effects of MB07811 on other lipid markers compared to placebo | 12 weeks
Assess the safety and tolerability of MB07811 | after 12 weeks of treatment and during off-drug phase

CONTACTS AND LOCATIONS:
Overall Officials: Trish Novak, Ph.D., Study Director — Metabasis Therapeutics, Inc.
Locations (11):
- United States (11):
  - Scripps Clinic, Clinical Research, San Diego, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University Clinical Research, Pembroke Pines, Florida
  - Radiant Research, Chicago, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Commonwealth Biomedical Research, Madisonville, Kentucky
  - Troy Internal Medicine, Troy, Michigan
  - Coastal Carolina Research Center, Inc., Goose Creek, South Carolina
  - Research Across America, Dallas, Texas
  - National Clinical Research - Norfolk, Norfolk, Virginia
  - National Clinical Research, Richmond, Virginia